CLINICAL TRIAL: NCT05693038
Title: Brachial Plexus Injury After Prone Positioning in Intensive Care Unit: a Prospective Observational Study
Brief Title: Brachial Plexus Injury After Prone Positioning
Acronym: BPX
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Principal Investigator, Filippo Binda, Principal Investigator, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Other Study IDs: 6057
Record Dates: First submitted 2022-12-29; First posted 2023-01-20 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Brachial Plexus Injury; Nerve Compression
Keywords: Prone Position; Brachial Plexus; Respiratory Distress Syndrome; Intensive Care Unit; Swimmer position
MeSH Terms: conditions — Neuroma; Respiratory Distress Syndrome | interventions — Electromyography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Electromyography — Electromyography (EMG) monitoring will be performed, using the instrumentation available (Nemus 2, EB Neuro, Italy), to evaluate the occurrence of brachial plexus injury (BPI). EMG will be performed at the end of each pronation cycle. To rule out BPI at ICU admission, an EMG will be performed within two hours from the first pronation maneuver. Particularly, somatosensory evoked potential (SSEP) and sensory action potential (SAP) will be obtained from radial, ulnar, median and sural nerves. In case patients are awake, compound muscle action potential (CMAP) will be obtained as well.
Diagnostic Test: Muscle strength measurement — Muscle strength measure willl be assessed at ICU discharge using hand-held dynamometer.

SUMMARY:
The goal of this prospective observational study is to estimate the prevalence of brachial plexus injury after prone positioning in patients with ARDS and to evaluate the safety of swimmer position. The main questions it aims to answer are:

* Could arm positioning during pronation play a role in the development of any nerve injury at the brachial plexus level?
* Is swimmer position safe when adopted during prone positioning?

Participants will be studied at selective time points using EMG assessment.

DETAILED DESCRIPTION:
Prone positioning will be performed according to the current guidelines. Particularly, face and limbs will be placed according to the "swimmer position", ensuring the face position in the direction of ventilator and limbs (one arm above head and opposite arm at side) positioned as to prevent abnormal extension or flexion against the shoulders and elbows. Patients will lie on low air loss pressure mattresses, thus avoiding the utilization of any thoraco-pelvic supports, which are not recommended. Electromyography (EMG) will be performed to evaluate the occurrence of brachial plexus injury (BPI).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Admission to ICU for severe ARDS
* Administration of sedation and neuromuscular blocking agents
* Presence of endotracheal intubation and mechanical ventilation
* Use of prone positioning to treat hypoxemia

Exclusion Criteria:

* Extracorporeal membrane oxygenation
* Prone positioning performed in other centers
* Prone positioning contraindications
* Neurodegenerative disorders
* Previous known brachial plexus injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted in the ICU with severe ARDS, also secondary to pulmonary involvement of COVID-19, receiving invasive mechanical ventilation and requiring prone positioning to treat hypoxemia, as decided by the medical team.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2022-04-06 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with signs of brachial plexus injury (BPI) | EMG will be perform at the end of the every cycle of prone positioning (each cycle is 16 hours on average) and within 24 hours before ICU discharge
  Signs of BPI are the presence of (almost one of four EMG results):
  * Somatosensory Evoked Potential N20 latency of radial nerve and ulnar nerve > 10% compared to baseline
  * Somatosensory Evoked Potential N20 amplitude of radial nerve and ulnar nerve < 50% compared to baseline
  * Sensory Action Potential amplitude of radial nerve, ulnar nerve and median nerve < 50% compared to baseline
  * Compound Motor Action Potential amplitude of ulnar and median nerve < 50% compared to normative data (assessed before ICU discharge)

SECONDARY OUTCOMES:
Safety of swimmer position adopted | The safety of the swimmer position will be evaluated within 24 hours before ICU discharge
  The safety is defined in terms of:
  * number of patients with adverse events during prone positioning
  * number of patients with pressure ulcers after prone positioning
  * number of patients with ocular damage after prone positioning
  * number of patients with auricle damage after prone positioning

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bamford P, Denmade C, Newmarch C, Shirley P, Singer B, Webb S, et al. Guidance For Prone Positioning in Adult Critical Care. Intensive Care Soc. 2019;1-39.
- [Background] Chiumello D, Cressoni M, Racagni M, Landi L, Li Bassi G, Polli F, Carlesso E, Gattinoni L. Effects of thoraco-pelvic supports during prone position in patients with acute lung injury/acute respiratory distress syndrome: a physiological study. Crit Care. 2006;10(3):R87. doi: 10.1186/cc4933. Epub 2006 Jun 8. PMID 16764731